CLINICAL TRIAL: NCT04420299
Title: A Randomized, Single-blind Study With a Parallel Control Group on the Efficacy and Safety of Bemiparin at Therapeutic Dose vs. Prophylactic Dose in Patients Hospitalized for COVID-19
Brief Title: Clinical Trial on the Efficacy and Safety of Bemiparin in Patients Hospitalized Because of COVID-19
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Lack of funding of the non-commercial sponsor to extend recruitment and reach the target number of patients specified in the protocol.
Sponsor: Fundación de investigación HM (Other)
Collaborators: Syntax for Science, S.L (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: BEMICOVID-19; 2020-001548-24 (EudraCT Number)
Record Dates: First submitted 2020-06-05; First posted 2020-06-09 (Actual); Last update posted 2022-06-07 (Actual); Status verified 2022-06

CONDITIONS: Covid-19
Keywords: covid-19; immunothrombosis; d-dimer
MeSH Terms: conditions — COVID-19; Thromboinflammation | interventions — bemiparin

STUDY DESIGN:
Intervention Model Description: randomized, single-blind, parallel control group
Who Masked: Participant
Masking Description: Subjects will be blinded to the dosing regimen (treatment dose or prophylactic dose).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental - therapeutic bemiparin dose (Experimental): Sub-cutaneous dose of bemiparin at therapeutic dose for 10 days
  Interventions: Drug: Bemiparin
- Control - prophylactic bemiparin dose (Experimental): Sub-cutaneous dose of bemiparin at prophilactic dose for 10 days
  Interventions: Drug: Bemiparin

INTERVENTIONS:
Drug: Bemiparin — Bemiparin at therapeutic dose for 10 days
  Other Names: Therapeutic dose
  Arms: Experimental - therapeutic bemiparin dose
Drug: Bemiparin — Bemiparin at prophylactic dose for 10 days
  Other Names: Prophylactic dose
  Arms: Control - prophylactic bemiparin dose

SUMMARY:
The 2019 coronavirus disease (Covid-19) is a new disease caused by the SARS-CoV2 virus of which many things are not yet known. Among others, there is a need to define the best therapeutic strategy to treat Covid-19, improving patients survival and reducing complications in its management, for which many different types of treatments are being tested.

The drug being tested in this clinical trial is called bemiparin. Bemiparin is a drug authorized as a prevention and as a treatment for deep vein thrombosis (blood clots in one or more veins, generally in the legs) and venous thromboembolism (when the clot can detach and lodge in other organs such as the lungs). Covid-19 patients have been shown to be at increased risk of developing clotting problems such as those described above.

In this context, this clinical trial is being carried out to find out if certain doses of bemiparin can contribute to better management of the disease.

ELIGIBILITY:
Inclusion Criteria:

1. Informed consent.
2. Age of 18 years or more.
3. Patient with suspected COVID-19 and who meets hospitalization criteria.
4. D-dimer> 500 ng / ml.
5. Clinical characteristics highly compatible with SARS-CoV-2 infection and confirmation by RT-qPCR at baseline or in the second sample in case of a first negative test and clinical suspicion remains.
6. Patient admitted to hospital

Exclusion Criteria:

1. ICU admission criteria.
2. Need for invasive or not invasive mechanical ventilation
3. Pregnancy.
4. Creatine clearance <30 ml / min (Cockroft-Gault).
5. Severe liver or pancreatic function disorder.
6. Acute bacterial endocarditis and slow endocarditis.
7. Patient previously anticoagulated (although it is allowed to have received heparin at a previous low dose without time limit).
8. Patient with high hemorrhagic risk due to previous medical-surgical history.
9. Severe thrombocytopenia (<80,000 platelets/ mm3) or known history of heparin-induced thrombocytopenia.
10. Active bleeding or increased risk of bleeding from haemostasis disorders or from organic lesions that are liable to bleed (eg, active peptic ulcer, hemorrhagic stroke, aneurysms, or brain malignancies).
11. Damage or surgical interventions in the central nervous system, eyes and ears that have taken place in the last 2 months.
12. Simultaneous participation in another clinical trial that could have a conflictive interaction with what it is intended to evaluate.
13. Any situation that in the opinion of the researcher could interfere with the treatment or with the evolution of the patient.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 81 (Actual)
Dates: Start 2020-06-04 (Actual); Primary Completion 2021-06-08 (Actual); Study Completion 2021-06-08 (Actual)

PRIMARY OUTCOMES:
Proportion of patients that worsen | Day 10 +/- 1
  Combined worsening variable. Presence of any of the following will be considered worseing:
  1. Death.
  2. ICU admission.
  3. Need for either non-invasive or invasive mechanical ventilation.
  4. Progression to moderate / severe respiratory distress syndrome according to objective criteria (Berlin definition).
  5. Venous thromboembolism (deep vein thrombosis or pulmonary embolism) or arterial (acute myocardial infarction or stroke).

SECONDARY OUTCOMES:
Mortality from any cause at day 28 | Day 28
  Mortality from any cause
Proportion of subjects that requires admission to the ICU | From study start to day 28
  Proportion of subjects that requires admission to the ICU
Proportion of subjects requiring non-invasive mechanical ventilation | From study start to day 28
  Proportion of subjects requiring non-invasive mechanical ventilation
Proportion of subjects requiring invasive mechanical ventilation. | From study start to day 28
  Proportion of subjects requiring invasive mechanical ventilation.
Proportion of subjects with some organ failure | From study start to day 28
  Proportion of subjects with some organ failure
Proportion of patients who have modified their oxygen therapy requirements between treatment assessment visit and baseline | From study start to day 28
  Proportion of patients who have modified their oxygen therapy requirements between treatment assessment visit and baseline
Proportion of subjects with pathological angioTAC | At day 10 +/-1
  Proportion of subjects with pathological angioTAC at day 10 +/-1
Proportion of subjects with improvement in chest radiography | At day 10 +/-1
  Proportion of subjects with improvement in chest radiography
Proportion and median hospital discharge between patients in both groups. | From study start to day 28
  Proportion and median hospital discharge between patients in both groups.
Titration score | From study start to day 28
  Titration score
Ferritin score | From study start to day 28
  Ferritin score
D-dimer modification score | From study start to day 28
  D-dimer modification score
Adverse events (total and serious). | From study start to day 28
  Adverse events (total and serious)
Related adverse events (total and serious). | From study start to day 28
  Related adverse events (total and serious).
Clinically relevant major and non major hemorrhages. | From study start to day 28
  Clinically relevant major and non major hemorrhages.

CONTACTS AND LOCATIONS:
Overall Officials: Antonio Cubillo, MD, Study Director — Director
Locations (2):
- Spain (2):
  - Hospital Universitario HM Montepríncipe, Boadilla del Monte, Madrid
  - Hospital Universitario HM Puerta del Sur, Móstoles, Madrid

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Flumignan RL, Civile VT, Tinoco JDS, Pascoal PI, Areias LL, Matar CF, Tendal B, Trevisani VF, Atallah AN, Nakano LC. Anticoagulants for people hospitalised with COVID-19. Cochrane Database Syst Rev. 2022 Mar 4;3(3):CD013739. doi: 10.1002/14651858.CD013739.pub2. PMID 35244208